CLINICAL TRIAL: NCT01929408
Title: Feasibility and Outcomes of Allogeneic Hematopoietic Cell Transplantation (HCT) Compared to Conventional Therapy for Older and Medically Infirm Patients Diagnosed With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes: A Prospective Observational Study
Brief Title: Feasibility and Outcomes of Allogeneic HCT Compared to Chemotherapy in Older AML Patients
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 2368.00; RSG-13-084-01-CPHPS (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2013-08-14; First posted 2013-08-28 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare treatment methods and outcomes of patients diagnosed with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
This is a prospective multicenter observational study in a Consortium of collaborating institutions investigating how often older and medically infirm patients who are diagnosed with Acute Myeloid Leukemia (AML) or high-risk myelodysplastic syndromes (MDS) and treated with induction chemotherapy undergo allogeneic HCT. Investigators will look at the rate of undergoing allogeneic HCT among older and medically infirm AML and high-risk MDS patients compared to younger and relatively healthier patients. Investigators will also compare the characteristics and outcomes of patients who did versus did not proceed to allogeneic HCT. A number of outcomes will be assessed including mortality, morbidity, and quality of life (QOL). Baseline information will be collected on different domains of QOL, geriatric assessment, health status measures, AML features, and socioeconomic status. Information will help physicians and patients to decide on best treatment choices for AML and high-risk MDS in older and medically infirm patients.

ELIGIBILITY:
Inclusion Criteria

Patients with new diagnoses of non-M3 AML or high-risk MDS, myeloproliferative neoplasms (MPN), or myelofibrosis (MF) (showing 10% or more blasts in bone marrow) who:

* Present for an AML-like treatment that could plausibly produce a complete remission (CR); for example intensive induction chemotherapy, low dose single agent chemotherapy, hypomethylation agent, or a similar therapy
* Possibility to retrieve follow-up records from the collaborating institution or treating primary care physician
* Patients with primary refractory or first relapse presenting for salvage chemotherapy will be allowed
* Patients of 18 years of age or older, and are being treated by the adult AML service.
* Able to speak and read English.
* Willing and able to provide informed consent.

Exclusion Criteria

* Patients of ≤17 years of age or who are 18 or older and receive treatment under the pediatric AML service.
* Patients older than 80 years
* Patients with <6 months projected survival due to active second malignancy or other medical problem.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include non-M3 AML (including first relapsed and primary refractory AML) and high-risk MDS, MPN, and MF adult patients considered for chemotherapy at FHCRC and the Seattle Cancer Care Alliance Network and other Core institutions (Stanford School of Medicine, Cleveland Clinic, Northwestern University, University of Utah, University of Pennsylvania, Washington University in St. Louis, Roswell Park Cancer Institute, Hackensack University, University of Maryland, and Duke University).
Sampling Method: Non-Probability Sample
Enrollment: 703 (Actual)
Dates: Start 2013-07-19 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sorror, MD, MSc, Principal Investigator — Associate Member, Fred Hutch; Associate Professor of Medicine, UW
Locations (12):
- United States (12):
  - Stanford Cancer Institute, Stanford, California
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - The John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - SCCA Network Clinics, Seattle, Washington

REFERENCES:
- [Derived] Sorror ML, Gooley TA, Storer BE, Gerds AT, Sekeres MA, Medeiros BC, Wang ES, Shami PJ, Adekola K, Luger S, Baer MR, Rizzieri DA, Wildes TM, Koprivnikar J, Smith J, Garrison M, Kojouri K, Schuler TA, Leisenring WM, Onstad LE, Becker PS, McCune JS, Lee SJ, Sandmaier BM, Appelbaum FR, Estey EH. An 8-year pragmatic observation evaluation of the benefits of allogeneic HCT in older and medically infirm patients with AML. Blood. 2023 Jan 19;141(3):295-308. doi: 10.1182/blood.2022016916. PMID 36260765
- [Derived] Sorror ML, Storer BE, Fathi AT, Brunner A, Gerds AT, Sekeres MA, Mukherjee S, Medeiros BC, Wang ES, Vachhani P, Shami PJ, Pena E, Elsawy M, Adekola K, Luger S, Baer MR, Rizzieri D, Wildes TM, Koprivnikar J, Smith J, Garrison M, Kojouri K, Leisenring W, Onstad L, Nyland JE, Becker PS, McCune JS, Lee SJ, Sandmaier BM, Appelbaum FR, Estey EH. Multisite 11-year experience of less-intensive vs intensive therapies in acute myeloid leukemia. Blood. 2021 Aug 5;138(5):387-400. doi: 10.1182/blood.2020008812. PMID 34351368

RESULTS

PARTICIPANT FLOW:
Groups:
- Acute Myeloid Leukemia (AML) & Myelodysplastic Syndrome (MDS): All patients starting induction therapy for newly diagnosed AML or advanced MDS and followed over time
Period: Overall Study
Arm/Group | Acute Myeloid Leukemia (AML) & Myelodysplastic Syndrome (MDS)
Started (Number Ss enrolled) | 703
Completed (Total Ss with analyzable data. Incomplete follow-up data could still be included in analyses.) | 695
Not Completed | 8
Not completed — received HCT as initial treatment | 8

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients enrolled on the study for treatment of their Acute Myeloid Leukemia (AML) or high-risk Myelodysplastic Syndrome (MDS) disease.
Arm/Group | All Patients
Number analyzed (Participants) | 703
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 436
  >=65 years | 267
Age, Continuous [Median (Full Range); unit: years] | 62 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304
  Male | 399
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 662
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 13
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 41
  White | 608
  More than one race | 3
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 703

OUTCOME MEASURES:

1. Primary Outcome: Percentage Analyzed Participants Receiving Hematopoietic Stem Cell Transplantation (HCT)
Description: Percentage analyzed participants receiving HCT
Time Frame: 1 year after starting induction
Measure: Number; unit: % participants
Groups:
- All Patients: All eligible patients enrolled on the study for treatment of their Acute Myeloid Leukemia (AML) or high-risk Myelodysplastic Syndrome (MDS) disease.
Arm/Group | All Patients
Number analyzed (Participants) | 695
% participants | 44.7

2. Secondary Outcome: Percentage Analyzed Participants Without HCT and Deceased
Description: Percentage analyzed participants without HCT and Deceased
Time Frame: 1 year after starting induction
Measure: Number; unit: % participants
Arm/Group | All Patients
Number analyzed (Participants) | 695
% participants | 32.7

ADVERSE EVENTS:
Time Frame: 1 year after starting induction
Description: Adverse events did not occur as a direct result of this observational study
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 309/695
Serious Adverse Events (participants affected / at risk) | 0/695
Other Adverse Events (participants affected / at risk) | 0/695

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT01929408/Prot_SAP_000.pdf